CLINICAL TRIAL: NCT02304484
Title: A Multicenter, Open-label Extension (OLE) Study to Assess the Long-term Safety and Efficacy of Evolocumab
Brief Title: Open-label Extension (OLE) Study to Assess Safety and Efficacy of Evolocumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140128; 2014-001524-30 (EudraCT Number)
Record Dates: First submitted 2014-10-07; First posted 2014-12-02 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Evolocumab (Experimental): Participants received 420 mg evolocumab once a month for up to 2 years.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection once a month
  Other Names: AMG 145; Repatha

SUMMARY:
The purpose of this study was to characterize the safety and tolerability of long-term administration of evolocumab in adults with known coronary artery disease and hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Completed week 80 of study 20120153 (NCT01813422).

Exclusion Criteria:

* Did not complete investigational product in the 20120153 parent study
* Have an unstable medical condition, in the judgment of the investigator
* Known sensitivity to any of the products to be administered during dosing
* Currently enrolled in another investigational device or drug study (excluding evolocumab (AMG 145) parent study), or less than 30 days since ending another investigational device or drug study(s),or receiving other investigational agent(s)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (115):
- United States (24):
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Long Beach, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Jacksonville, Florida
  - Research Site, Munster, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Bay City, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Ridgewood, New Jersey
  - Research Site, Fargo, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Dallas, Texas
  - Research Site, Wichita Falls, Texas
- Argentina (3):
  - Research Site, La Plata, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Córdoba
- Australia (9):
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Epping, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Nedlands, Western Australia
- Belgium (5):
  - Research Site, Antwerp
  - Research Site, Edegem
  - Research Site, Genk
  - Research Site, Hasselt
  - Research Site, Lodelinsart
- Brazil (2):
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, Temuco, Cautín, Chile
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Zlín
- France (5):
  - Research Site, Besançon
  - Research Site, Chambray-lès-Tours
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Pessac
- Research Site, Essen, Germany
- Greece (2):
  - Research Site, Athens
  - Research Site, Heraklion
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Research Site, Reykjavik, Iceland
- Research Site, Galway, Ireland
- Israel (2):
  - Research Site, Hadera
  - Research Site, Jerusalem
- Italy (4):
  - Research Site, Novara
  - Research Site, Rozzano MI
  - Research Site, Sesto San Giovanni (MI)
  - Research Site, Torino
- Malaysia (2):
  - Research Site, Kuantan, Pahang
  - Research Site, George Town
- Mexico (4):
  - Research Site, Guadalajara, Jalisco
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Culiacán, Sinaloa
  - Research Site, Aguascalientes
- Netherlands (8):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Leeuwarden
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Zwolle
- Research Site, Oslo, Norway
- Poland (5):
  - Research Site, Chrzanów
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Kemerovo
  - Research Site, Moscow
- South Africa (3):
  - Research Site, Centurion, Gauteng
  - Research Site, Sunninghill, Gauteng
  - Research Site, Kuils River, Western Cape
- South Korea (3):
  - Research Site, Daejeon
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Seoul
- Spain (5):
  - Research Site, Málaga, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Madrid
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- Research Site, Geneva, Switzerland
- Research Site, New Taipei City, Taiwan
- Research Site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 126 centers in 29 countries in the regions of Europe, North America, Asia Pacific, and Latin America. Participants were enrolled from 24 November 2014 to 31 August 2016.
Pre-assignment Details: Participants who successfully completed week 80 of the parent Study 20120153 (NCT01813422) and did not discontinue study drug in the parent study for any reason were eligible for this study. All participants received open-label evolocumab.
Period: Overall Study
Arm/Group | Evolocumab
Started | 770
Completed | 745
Not Completed | 25
Not completed — Death | 9
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants. Baseline is defined as parent study 20120153 baseline.
Arm/Group | Evolocumab
Number analyzed (Participants) | 770
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.8)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 536
  ≥ 65 years | 234
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 568
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 732
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 19
  Black or African American | 5
  Native Hawaiian or Other Pacific Islander | 1
  White | 729
  Multiple | 11
  Other | 4
Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Baseline is defined as parent study 20120153 baseline.
  mg/dL | 92.2 (27.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event (AE) was graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 criteria, where Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe or medically significant AE, Grade 4 = Life-threatening consequences, and Grade 5 = death related to AE.
  An adverse device effect was defined as any adverse event related to the use of a medical device (autoinjector/pen or automated mini doser [AMD]), including but not limited to, AEs resulting from insufficient or inadequate Instructions for Use, AEs resulting from any malfunction of the device, or AEs resulting from use error or from intentional misuse of the device.
Time Frame: From first dose of evolocumab up to 30 days after the last dose, or end of study, whichever was earlier, up to 108 weeks.
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Evolocumab
Number analyzed (Participants) | 770
Participants
  Any adverse event | 526
  Adverse events ≥ Grade 2 | 415
  Adverse events ≥ Grade 3 | 206
  Adverse events ≥ Grade 4 | 38
  Serious adverse events | 153
  AEs leading to discontinuation of evolocumab | 14
  Fatal adverse events | 6
  Device-related adverse events | 12
  Device-related adverse events ≥ Grade 2 | 2
  Device-related adverse events ≥ Grade 3 | 1
  Device-related adverse events ≥ Grade 4 | 0
  Serious device-related adverse events | 0

2. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: Baseline (of study 20120153) and weeks 0, 4, 12, 24, 36, 48, 52, 76, and 104 of study 20140128
Population: Enrolled participants with available data at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Evolocumab
Number analyzed (Participants) | 770
percent change
  Percent change from baseline to week 0: number analyzed (Participants) | 751
  Percent change from baseline to week 0 | -21.52 (40.49)
  Percent change from baseline to week 4: number analyzed (Participants) | 752
  Percent change from baseline to week 4 | -57.23 (22.19)
  Percent change from baseline to week 12: number analyzed (Participants) | 746
  Percent change from baseline to week 12 | -58.54 (25.60)
  Percent change from baseline to week 24: number analyzed (Participants) | 747
  Percent change from baseline to week 24 | -55.26 (28.51)
  Percent change from baseline to week 36: number analyzed (Participants) | 738
  Percent change from baseline to week 36 | -51.72 (30.34)
  Percent change from baseline to week 48: number analyzed (Participants) | 709
  Percent change from baseline to week 48 | -53.65 (28.72)
  Percent change from baseline to week 52: number analyzed (Participants) | 725
  Percent change from baseline to week 52 | -51.30 (28.48)
  Percent change from baseline to week 76: number analyzed (Participants) | 722
  Percent change from baseline to week 76 | -51.73 (32.49)
  Percent change from baseline to week 104: number analyzed (Participants) | 607
  Percent change from baseline to week 104 | -47.94 (36.49)

ADVERSE EVENTS:
Time Frame: Total deaths are reported from the 1st dose of evolocumab up to the end of study; adverse events are reported from the 1st dose of evolocumab up to 30 days after the last dose of study drug or end of study, whichever was earlier. The median (minimum, maximum) duration of treatment was 23.7 (0.4, 24.6) months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Evolocumab
All-Cause Mortality (participants affected / at risk) | 9/770
Serious Adverse Events (participants affected / at risk) | 153/770
Other Adverse Events (participants affected / at risk) | 49/770
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=770)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 13
Angina unstable (Cardiac disorders) | 5
Arteriospasm coronary (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 4
Coronary artery stenosis (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Cataract (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 4
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 6
Sudden death (General disorders) | 1
Vascular stent occlusion (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 3
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1
Contrast media reaction (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 2
Bacterial colitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Staphylococcal osteomyelitis (Infections and infestations) | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Anticoagulation drug level above therapeutic (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to urinary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Cervical radiculopathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 2
Device loosening (Product Issues) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=770)
Hypertension (Vascular disorders) | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02304484/SAP_000.pdf
  • Study Protocol (2014-12-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02304484/Prot_001.pdf